CLINICAL TRIAL: NCT03321591
Title: Maternal Cognitive Function and Neurobehavioral Development of Underprivileged Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Dhaka (Other)
Responsible Party: Principal Investigator, Abu Yusuf Mahmud, Principal Investigator, University of Dhaka
Other Study IDs: 89/2015-16
Record Dates: First submitted 2017-10-13; First posted 2017-10-25 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is estimated that over 200 million children under 5 years of age in developing countries are not attaining their developmental potential (e.g., neurobehavioral development) primarily because of poverty and associated health, nutritional deficiencies, and unstimulating home environment. Child's Neurobehavioral development consists of several interdependent domains of sensory-motor, cognitive-language, and social-emotional function. Experiences in the first few years of life are of particular importance because vital development occurs during this period. Early under nutrition, iron-deficiency, environmental toxins, stress, and poor stimulation and social interaction can affect brain structure and function. Stunting, inadequate cognitive stimulation, iodine deficiency, and iron deficiency anemia are identified as key risk factors, where the need for cognitive intervention is urgent, that prevent millions of young children from fulfilling their developmental potential and neurobehavioral development. It is clear that underprivileged children require not only good health, nutrition, and wealth but also supportive and caring environments and cognitive stimulation for their optimum neurobehavioral development as in the case of Bangladesh. Cognitive function and self-esteem of mothers is crucial for having the optimum outcome from intervention. However, little is known regarding the importance of mother's cognitive ability influencing different domains of her children's neurobehavioral development. This is how, the investigators plan to measure the maternal cognitive function and to assess the neurobehavioral development of underprivileged children. The investigators will enroll 200 mothers and children as a sample of the present study. Bayley Scales of Infant and Toddler Development will be used along with other interview scales.

DETAILED DESCRIPTION:
Child development consists of several interdependent domains of sensory-motor, cognitive-language, and social-emotional function. Children's development is affected by psychosocial and biological factors through changes in brain structure and function, and behavioral changes. Experiences in the first few years of life are of particular importance because vital development occurs in all the domains during this period, and the interaction between early environments and genetics influences this development and human behavior. The brain growth occurs rapidly through neurogenesis, axonal and dendritic proliferation, synaptogenesis, cell death, synaptic pruning, myelination, and gliogenesis. Brain development can be modified by the quality of the environment. Independent animal research suggests that early under nutrition, iron-deficiency, environmental toxins, stress, and poor stimulation and social interaction can affect brain structure and function. In both humans and animals, variations in the quality of maternal care, a part of home environment, can yield changes in stress reactivity, anxiety, and memory function in the offspring. In later childhood the affected children will subsequently have lower levels of cognition and education. It is mentionable that remarkable recovery is often possible with early intervention through more nurturing environment with adequate stimulation, despite the vulnerability of the brain to early insult.

Stunting, inadequate cognitive stimulation, iodine deficiency, and iron deficiency anemia are identified as key risk factors, where the need for intervention is urgent, that prevent millions of young children from fulfilling their developmental potential. In low-income and middle-income countries, 34% of children younger than 5 years have linear growth retardation or stunting resulted from poor nutrition often accelerated by infectious diseases. It is reported that patterns of growth retardation are identical across countries. Although the vacillation in growth starts in utero or in the first 12-18 months, continue to around 40 months, but most children having stunting remain stunted through to adulthood. On the other hand, poverty and stunting are identified for indicators of poor development because the researchers represent different types of biological and psychosocial risks. Poverty is related to inadequate food, and poor sanitation and hygiene that increase infections and stunting in children. Poverty is also connected to poor maternal education, increased maternal stress and depression, and deficient stimulation in the home. All these factors deleteriously affect child development which, in turn, produces poor school achievement, which is further worsened by poor family support. Risk factors associated with poverty frequently happen together, and degree of development becomes lower with the number of risks factors. Deficits in child development are often occurred in infancy and increase further with age. Several longitudinal studies have found substantial association between socioeconomic status and parental wealth at birth, and cognitive attainment. Poverty and sociocultural background increase children's exposure to psychosocial risks that influence development through behavioral changes.

Parenting factors like cognitive stimulation or learning opportunities facilitates early cognitive development. Several studies examined the effect of stimulation or intervention on children from developing countries, including children living in poverty, which strongly supports the importance of early cognitive intervention for facilitating better cognitive and non-cognitive outcomes. Research revealed three aspects of parenting associated to young children's cognitive and social-emotional competence: cognitive stimulation, caregiver sensitivity and responsiveness to the child, and caregiver affect (National Research Council and Institute of Medicine. Regarding maternal sensitivity and responsivity several researches reported that these factors are associated with more secure infant attachment and higher cognitive ability respectively. Appropriate caregiver-child interactions facilitate early social-emotional development and learning materials promote age-appropriate language and problem-solving skills. These factors discussed above are the part of maternal cognitive function which implies that there might be a link between factors evolved from maternal cognitive state and child development. Showed that maternal cognitive ability works as an important factor in progressing children's height, even after controlling for child's age and gender, parental age, mother's and father's years of schooling and mother's height.

It is worth mentioning that substantial improvement in development is unlikely to be made without also increasing early learning opportunities, though there has been recent attention to the effect of nutrition on development. Non-US intervention studies showed that cognitive benefits were better in case of interventions having stimulation and education components compared with those involving nutrition or economic assistance only. In Bangladesh, research revealed that almost 60% children are exposed to risk of insufficient development caused by high prevalence of LBW (22%), stunting (41%), and poverty (43%), and lack of early stimulation due to low parental knowledge. Most of the data from developing countries including Bangladesh mainly focused on cognitive and motor outcome with less emphasis on maternal cognitive ability. This is why, in addition to the existing information, the investigators need to assess maternal cognitive ability and neurobehavioral development in order to prepare appropriate intervention particularly for disadvantaged children living in poverty in Bangladesh.

It is clear from the previous studies on poor populations that disadvantaged children require not only good health, nutrition, and wealth but also supportive and caring environments at home and cognitive stimulation in order to achieve their developmental potential as in the case of Bangladesh. According to Lancet review, most disadvantaged children get the maximum benefit of intervention. Cognitive function of parents, especially mothers, is crucial for having the optimum outcome from intervention. However, little is known regarding the importance of mother's cognitive functioning influencing different domains of her young children's neurobehavioral developmental outcome mediated by parenting, particularly who are from disadvantageous community in Bangladesh, residing in poverty. The investigators know of no other study, however, that directly emphasizes maternal cognitive function on different domains of development of disadvantaged children in Bangladesh.

The investigators, therefore, plan to examine the association of disadvantaged children's neurobehavioral development i.e., communication, motor skills, problem-solving, and personal-social skills and mother's cognitive function.

Hypothesis: Mothers with better cognitive function will have children with better neurobehavioral development.

Objectives: The specific objectives of the study are (a) to measure the maternal cognitive function, (b) to assess the neurobehavioral development of children.

A total of 200 mother-child will participate in the study. Data will be collected by the researchers or his representatives. Age range of children will range from 12-42 months residing in the slum area located in the city of Dhaka.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12-42 months on enrolment
* Sex: both male and female
* Living within 30 minutes distance from the center where the test takes
* place
* Nutritional status: weight-for-age z score (WAZ)>-3SD
* Consent: written consent provided by parents

Exclusion Criteria:

* Developmental anomalies,
* Known chronic illnesses like epilepsy, tuberculosis, mental retardation
* Twins and multiple births,
* Parents not consenting

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The sample (mothers & children) is collecting from the underprivileged population
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Cognitive, Language and Motor Composite Score | 6 months
  The outcomes are measured on Bayley Scales of Infant and Toddler Development, (3rd Edition). It measures three domains of child's development viz cognitive, language (receptive communication & expressive communication), and motor (fine motor & gross motor). The score of these three domains (or subscales) is calculated separately by adding up item score. Each item will get either 1 or 0. How many items is approached is dependent on child's age. Children having 16 days to 42.5 months are divided into 17 age groups having different starting point for item administration. Cognitive subscale has 91 items. Minimum and maximum scores will be 0 to 91. Language scale is comprised of receptive and expressive communication subtest. Total items of receptive and expressive subtests are 49 and 48 respectively & ranges will be 0-49 and 0-48. Gross and fine motor have 66 & 72 items and ranges 0-66 & 0-72. The higher the score the better the developmental outcome will be.
Maternal Cognitive Function Score | 6 months
  This outcome is measured on the mothers of children using The Bangla adaptation of Mini-Mental State Examination (BAMSE)
Behavior ratings | 6 months
  The outcome is observed using Wolke's behavior ratings during the administration of the Bayley Scales of Infant and Toddler Development .

SECONDARY OUTCOMES:
Child's Home environment observation | 6 months
  Child's home environment will be assessed using home observation measurement of the environment (HOME) scale. It measures the quality of the child's home environment and quality of cognitive stimulation & emotional support provided by a child's family. The scale is comprised of 36 items. Each item will receive either 0 or 1 score. Thus the range of total score is minimum 0 and maximum 36. The higher the score the better the child's home environment quality.
Parent child interactions | 6 months
  This outcome is measured by the bangla version of parenting scale. This is a 20-item measure of typical everyday events in parenting and parent-child interactions. This outcome will be obtained by the interviews with the mothers of the children. Each item has 4 response options ranging from 0 to 3. Thus range of total score will be 0 to 60. The higher the score the better the parenting will be.
Self-Esteem of mothers | 6 months
  This outcome is measured by the Bangla version of the Rosenberg self-esteem scale This is a 8-item scale having 5 response options which determines the self-esteem of mothers with interviews. Each item gets a score ranging from 0 to 4. Therefore, range of minimum and maximum total score is 0 to 32. The higher the score the strong the self-esteem.
Weight & height for Anthropometry measures | 6 months
  Children and mother's weight in kilograms and height in meters are measured using standard method. Then the weight and height will be combined to report BMI using standard technique
Mid Upper Arm Circumference (MUAC) | 6 months
  MUAC will be measured in meters by using tape to know the nutritional status
Head Circumference | 6 months
  Head circumference in meters of children will be measured by using tape for the growth status

CONTACTS AND LOCATIONS:
Overall Officials: MD. KAMAL UDDIN, PhD, Study Director — University of Dhaka
Locations (1):
- ICDDRB, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03321591/Prot_002.pdf
  • Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT03321591/SAP_003.pdf